CLINICAL TRIAL: NCT02246530
Title: Non-Surgical Treatment for Rotator-Cuff Tears Using Platelet-Rich-Plasma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prematurely due to inability to complete recruitment of subjects for each of the trial groups (treatment and control).
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Breanna Willeford, Resident Physician, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: F131231006
Record Dates: First submitted 2014-08-21; First posted 2014-09-22 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Partial Tear of Rotator Cuff; Tendinopathy of Rotator Cuff
MeSH Terms: interventions — Biological Products; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP injection into PTRCT (Active Comparator): Treatment - PRP injection
  Interventions: Procedure: PRP injection into PTRCT
- Subacromial steroid bursal injection (Active Comparator): Current standard of care for treatment of resistant partial thickness rotator cuff tears
  Interventions: Drug: Subacromial steroid bursal injection

INTERVENTIONS:
Procedure: PRP injection into PTRCT — Day of procedure, 60 cc blood draw will be taken for processing and isolation of PRP. PRP sample will be injected peri-tendinous / intra-tendinous area at location of the PTRCT under ultrasound guidance to ensure accurate placement at site of injury.
  PRP is an autologous blood product that is being re-injected into the same patient and is considered a non-invasive interventional procedure. PRP is classified as a procedure and not a drug.
  Other Names: Biologics
  Arms: PRP injection into PTRCT
Drug: Subacromial steroid bursal injection — Combination steroid (Celestone) and anesthetic drug (Lidocaine) will be injected into the patient's subacromial bursa via needle guidance of ultrasound
  Other Names: Procedure
  Arms: Subacromial steroid bursal injection

SUMMARY:
The goal of this project is to identify an effective and conservative approach to treating partial thickness rotator cuff tears (PTRCT) that otherwise would end with a surgical correction needed.

DETAILED DESCRIPTION:
Based off literature and clinical practice, the majority of rotator cuff tears continue to progress to surgical correction despite conservative measures. These include physical therapy, medication management and minimally invasive procedures such as subacromial bursa injections and intra-articular injections with steroids. Recently a popular treatment of common musculoskeletal injuries (including tendinopathies) has emerged throughout the US and has been utilized worldwide for many years with good empiric evidence known as Platelet-Rich Plasma (PRP) injections. In partnership with UAB Orthopedics and Radiology, the UAB Department of Physical Medicine and Rehabilitation aims to compare PRP to corticosteroid injections for patients with partial rotator cuff tears or tendinopathy. Outcome measures are ultrasound imaging, pain and disability over the course of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. subjects between ages 19 to 75, both male and female
2. radiologic imaging which can include either magnetic resonance imaging (MRI) or ultrasound (US) consistent with partial thickness rotator cuff tears of any degree except for full thickness tears
3. Failed a trial of physical therapy of at least 4 weeks

Exclusion Criteria:

1. Full thickness tears (well documented need for surgical correction)
2. sensory or neurologic complaint affecting the shoulder of interest
3. Coagulation disorder, platelet disorder
4. Pregnancy: Pregnancy test will be performed on women of childbearing age prior to their participation in the interventional portion of the study
5. Any major systemic illness such as ongoing infection or any condition that requires strict anti-platelet or anticoagulation therapy
6. Prior surgery to either cervical spine or shoulder
7. Active military
8. Injury part of worker compensation claim

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Breanna Willeford, DO, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Highlands, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from an outpatient Physical Medicine and Rehabilitation clinic at the University of Alabama. Each subject was given information regarding the study requirements and follow up obligations prior to enrollment and signed to complete based on their confidentiality agreement form.
Pre-assignment Details: Three subjects in this study were enrolled however prior to randomization in to their respective groups, they had a negative diagnostic ultrasound thus they were excluded from the study.
Groups:
- PRP Injection Into PTRCT: Treatment - PRP injection
  PRP injection into PTRCT: Day of procedure, 60 cc blood draw will be taken for processing and isolation of PRP. PRP sample will be injected peri-tendinous / intra-tendinous area at location of the PTRCT under ultrasound guidance to ensure accurate placement at site of injury.
  PRP is an autologous blood product that is being re-injected into the same patient and is considered a non-invasive interventional procedure. PRP is classified as a procedure and not a drug.
Period: Overall Study
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
Started | 9 | 2
Completed | 5 | 2
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 48.13 [28 to 62] | 57.5 [55 to 60] | 50 [28 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 11
SPADI (Shoulder Pain and Disability Index) Score [Mean (Full Range); unit: SPADI Score] — Comparing the questionnaire Shoulder Pain and Disability Index (SPADI) Scores pre-intervention in each group. The SPADI is a self-administered questionnaire that addressed pain and disability in functional activities. The raw score ranges from 0 (no pain or disability) to 130 (highest pain in each pain category and highest difficulty in each functional category). The SPADI Score is then calculated as a percentage (raw score divided by 130). Thus the final score is a range of 0% to 100%.
  SPADI Score | 43.69 [20.77 to 62.31] | 23.08 [21.54 to 24.62] | 37.80 [20.77 to 62.31]

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Ultrasound
Description: Comparing baseline diagnostic ultrasound for structural changes. An initial diagnostic ultrasound image was obtained to demonstrate a tear of the supraspinatus tendon, a key tendon of the rotator cuff. Once a tear of this tendon was confirmed, patient were delegated to one of the study arms and proceeded to the injection phase of the study.
  Two subject's data (within the PRP group) is incomplete as these subjects were lost to follow up and do not have completed 6 month follow up ultrasound imaging to review.
Time Frame: 6 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
Number analyzed (Participants) | 5 | 2
Participants
  Incomplete data (lost to follow up) | 1 | 0
  Number with improved (smaller) tear at follow up | 2 | 0
  Number with resolved tear at follow up | 2 | 2

2. Secondary Outcome: Shoulder Pain and Disability Index
Description: Comparing the questionnaire Shoulder Pain and Disability Index (SPADI) Scores to assess improvement after intervention. The SPADI is a self-administered questionnaire that addressed pain and disability in functional activities. The raw score ranges from 0 (no pain or disability) to 130 (highest pain in each pain category and highest difficulty in each functional category). The SPADI Score is then calculated as a percentage (raw score / 130). Thus, the final score is a range of 0% to 100%.
  In the PRP (platelet rich plasma injection) group we had 5 participants completed the study.
  2 participants in the control (corticosteroid injection) group completed the study.
Time Frame: Week 3 post procedure SPADI Scores for the control and treatment groups.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
Number analyzed (Participants) | 5 | 2
scores on a scale | 16.00 [2.31 to 54.62] | 18.08 [17.69 to 18.46]

3. Secondary Outcome: Shoulder Pain and Disability Index
Description: as for outcome 2
Time Frame: Week 6 post procedure SPADI Scores for the treatment and control groups.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
Number analyzed (Participants) | 5 | 2
scores on a scale | 8.00 [0 to 24.62] | 18.46 [15.38 to 21.54]

4. Secondary Outcome: Shoulder Pain and Disability Index
Description: as for outcome 2
Time Frame: 6 months post procedure SPADI scores for the treatment and control groups.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
Number analyzed (Participants) | 5 | 2
scores on a scale | 3.08 [0 to 4.62] | 7.31 [3.08 to 11.54]

ADVERSE EVENTS:
Time Frame: Patients were observed and monitored for adverse events up to 6 months post-procedure
Arm/Group | PRP Injection Into PTRCT | Subacromial Steroid Bursal Injection
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-07-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT02246530/Prot_000.pdf